CLINICAL TRIAL: NCT02641899
Title: A Phase 1, Fixed-Sequence, Open-label Study in Healthy Subjects to Estimate the Effects of ITCA 650 on Gastric Emptying and on the Absorption Pharmacokinetics of Each of 4 Commonly Studied Drug/Drug Interaction (DDI) Probe Compounds
Brief Title: Study of the Effects of ITCA 650 on Gastric Emptying and Interaction of ITCA 650 on 4 Commonly Studied Drugs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intarcia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ITCA 650-CLP-115
Record Dates: First submitted 2015-12-21; First posted 2015-12-30 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
Keywords: Adult; Male; Female; Volunteers
MeSH Terms: interventions — Exenatide; Acetaminophen; Atorvastatin; Lisinopril; Warfarin; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental Treatment (Experimental): ITCA 650 20/60 mcg/day Acetaminophen 1000 mg Atorvastatin 40 mg Lisinopril 20 mg Warfarin 25 mg Digoxin 0.5 mg
  Interventions: Drug: ITCA 650 20/60 mcg/day; Drug: Acetaminophen; Drug: Atorvastatin; Drug: Lisinopril; Drug: Warfarin; Drug: Digoxin

INTERVENTIONS:
Drug: ITCA 650 20/60 mcg/day — ITCA 650 osmotic mini pump delivering exenatide 20 mcg/day for 14 days, followed by ITCA 650 osmotic mini pump delivering exenatide 60 mcg/day.
Drug: Acetaminophen — Oral acetaminophen 1000 mg on Day 1 and Day 27
Drug: Atorvastatin — Oral atorvastatin 40 mg on Day 2 and Day 28
Drug: Lisinopril — Oral lisinopril 20 mg on Day 2 and Day 28
Drug: Warfarin — Oral warfarin 25 mg on Day 2 and Day 28
Drug: Digoxin — Oral digoxin 0.5 mg on Day 2 and Day 28

SUMMARY:
A Phase 1, Fixed-Sequence, Open-label Study in Healthy Subjects to Estimate the Effects of ITCA 650 on Gastric Emptying and on the Absorption Pharmacokinetics of Each of 4 Commonly Studied DDI Probe Compounds.

DETAILED DESCRIPTION:
Acetaminophen will be use to assess the effect of ITCA 650 on the rate of gastric emptying.

Interactions between ITCA 650 and the medications lisinopril, digoxin, atorvastatin, and warfarin will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 19 to 32 kg/m2.
* Glycosylated hemoglobin A1c (HbA1c )<6.5%.
* Normal renal function (eGFR ≥80 mL/min/1.73 m2).
* Women of child bearing potential - use of an additional adequate method of contraception during the study and until 1 additional menstrual cycle following the end-of-study (EOS) visit. Adequate methods of contraception for women of child bearing potential (WOCBP) include: mechanical products (ie, intrauterine device [IUD]-copper IUD); or barrier methods (eg, diaphragm, condoms, cervical cap) with spermicide.

Exclusion Criteria:

* History of type 1 or type 2 diabetes.
* History or evidence of myocardial infarction, coronary revascularization (coronary artery bypass grafting or percutaneous coronary intervention), unstable angina, or cerebrovascular accident or stroke.
* History of uncontrolled hypertension.
* History or evidence of acute or chronic pancreatitis.
* History of liver disease.
* History of medullary thyroid cancer or a personal or family history of multiple endocrine neoplasia type 2.
* Poor thyroid, liver, or renal function.
* Weight loss surgery or requires weight loss medications.
* History of malignancy (not including basal or squamous cell carcinoma of the skin with past 5 years). (Subjects who have been disease free for 5 years may be included.)
* History of active alcohol or substance abuse.
* Weekly consumption of more than 7 alcoholic beverages for females and 14 alcoholic beverages for males.
* Excessive in xanthine consumption (more than 5 cups of coffee or equivalent per day).
* Treatment with medications that affect GI motility.
* Any condition that would affect drug transit time or absorption (eg, gastrointestinal bypass surgery, partial or total gastrectomy, small bowel resection, chronic diarrhea, vagotomy, chronic gastroesophageal reflux disease, malabsorption, colostomy, Crohn's disease, ulcerative colitis, or celiac sprue).
* History of hypersensitivity to exenatide.
* Contraindications or warnings according to the specific label(s) for acetaminophen, atorvastatin, lisinopril, digoxin or warfarin therapy.
* Women that are pregnant, lactating, or planning to become pregnant.
* Concurrent use of anticoagulants, including daily low dose aspirin (81 mg).
* History of or positive results on screening tests for hepatitis B and/or hepatitis C and/or human immunodeficiency virus (HIV).
* Planned in-patient surgery, dental procedure, or hospitalization during the study.
* Prior or current treatment with any glucagon-like peptide-1 (GLP-1) receptor agonist (eg, Bydureon™, Byetta®, Victoza®, Tanzeum® or exogenous native GLP-1) or prior participation in an ITCA 650 clinical trial.
* Use or intended use of any drug or other product that inhibits or induces cytochrome P450 (CYP)1A2, CYP2C9, CYP2C19, or CYP3A4 within 14 days prior to the first dose of warfarin or ITCA650 or during the conduct of the study.
* History of thrombophlebitis, thromboembolic disorders, or deep vein thrombophlebitis.
* Fasting triglycerides above upper limit of normal at Screening.
* Any gastrointestinal complaints within 7 days prior to first dosing.
* Taking drugs or natural herbal supplements (such as albuterol, antacids, and St. John's Wort) with known interactions with atorvastatin, lisinopril, digoxin, or warfarin from within 7 days prior to Day 1 until EOS
* Consumed or unwilling to refrain from grapefruit, cranberries, grapefruit- or cranberry-containing products, or Seville oranges from within 7 days prior to Day 1 until EOS.
* Chronic use of analgesics, pain medication, or non-steroidal anti-inflammatory agents.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero to the last measurable concentration [AUC(0-last)]) of acetaminophen alone and in the presence of ITCA 650. | time zero to 10 weeks
Maximum plasma concentration ([Cmax]) of acetaminophen alone and in the presence of ITCA 650 | time zero to 10 weeks
Area under the concentration-time curve (AUC(0-last)) of atorvastatin, lisinopril, digoxin, R-warfarin, and S-warfarin each alone and in the presence of ITCA 650. | time zero to 10 weeks
Cmax of atorvastatin, lisinopril, digoxin, R-warfarin, and S-warfarin each alone and in the presence of ITCA 650. | time zero to 10 weeks

SECONDARY OUTCOMES:
Time to maximum plasma concentration (tmax) of acetaminophen | time zero to 10 weeks
tmax of atorvastatin, lisinopril, digoxin, R warfarin, and S-warfarin | time zero to 10 weeks
AUC(0-last) of orthohydroxy-atorvastatin and parahydroxy-atorvastatin | time zero to 10 weeks
Cmax of orthohydroxy-atorvastatin and parahydroxy-atorvastatin | time zero to 10 weeks
Maximum effect (Emax)from time zero to the last measurable concentration (AUEC(0-last)) of international normalized ratio (INR) of warfarin. | time zero to 10 weeks
Cmax of ITCA 650, 20 mcg/d and 60 mcg/d | within 8 hours after placement of ITCA 650
Treatment-emergent adverse events (TEAEs) including any events local to the placement site, clinical laboratory measurements, ECGs, vital signs and physical examinations. | time zero to 10 weeks
Tmax of orthohydroxy-atorvastatin and parahydroxy-atorvastatin | time zero to 10 weeks
Cmin of ITCA 650, 20 mcg/d and 60 mcg/d | time zero to 10 weeks
Tmax of ITCA 650, 20 mcg/d and 60 mcg/d | time zero to 10 weeks
Tmin of ITCA 650, 20 mcg/d and 60 mcg/d | zero to 10 weeks
Time of maximum effect (tEmax)from time zero to the last measurable concentration (AUEC(0-last)) of international normalized ratio (INR) of warfarin. | zero to 10 weeks
Area under the effect-time curve from time zero to the last measurable concentration (AUEC(0-last)) of international normalized ratio (INR) of warfarin. | zero to 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No